CLINICAL TRIAL: NCT06918899
Title: Identifying the Prevalence of Complex Post-Traumatic Stress Disorder in Trauma-Exposed Children and Adolescents and Examining Related Factors
Brief Title: Prevalence of Complex PTSD in Trauma-Exposed Children-Adolescents and Related Factors
Status: Recruiting | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Beyza Nur Karal, Research Assistant, MD, Istanbul University
Other Study IDs: 2025/82
Record Dates: First submitted 2025-03-20; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Complex Post-Traumatic Stress Disorder (CPTSD); Post-traumatic Stress Disorder (PTSD)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to assess the psychiatric evaluation of children and adolescents exposed to trauma in the outpatient clinic and to determine the prevalence of PTSD and Complex PTSD (CPTSD) diagnoses. Additionally, it aims to compare the clinical characteristics of children exposed to trauma who do not receive a PTSD diagnosis, those diagnosed with PTSD, and those diagnosed with CPTSD, as well as to examine the trauma history of their parents and the severity of their anxiety and depression. Furthermore, since there is no existing scale to assess CPTSD in children in our country, the study also aims to translate the International Trauma Questionnaire - Child and Adolescent Version into Turkish and evaluate its psychometric properties.

DETAILED DESCRIPTION:
The study will be conducted under the coordination of the Department of Child and Adolescent Psychiatry at Istanbul Faculty of Medicine. The sample will consist of children and adolescents who have been identified by their attending physician as having experienced trauma and have been referred to participate in the study at the Child and Adolescent Psychiatry outpatient clinic of Istanbul Faculty of Medicine.

Sample:

* Children and adolescents aged 7-18,
* Children and adolescents who have experienced trauma and applied to the Child and Adolescent Psychiatry outpatient clinic of Istanbul Faculty of Medicine,
* Children and/or parents with adequate literacy and Turkish language skills,
* Those without psychotic/manic symptoms or a diagnosis of autism spectrum disorder or intellectual disability in the child or parent during the interview,
* Volunteers who agree to participate in the study.

Researchers will explain the study to volunteer children and their families and present the Informed Consent Form to determine their willingness to participate.

Parents of eligible volunteers will complete the following assessments:

* Sociodemographic Data Form
* Hospital Anxiety and Depression Scale
* Advers Childhood Events Scale
* Positive Childhood Experiences Scale
* Strengths and Difficulties Questionnaire (Parent Form)

Volunteer children and adolescents will complete:

* International Trauma Questionnaire - Child and Adolescent Version
* Revised Children's Anxiety and Depression Scale
* Positive Childhood Experiences Scale
* (Adolescent/Child's Self Report) Responses to Stress Questionnaire (Peer Stress)

The clinician will conduct the following assessments:

* ICD-11-based clinical interview
* UCLA PTSD Reaction Index for DSM-5
* Children's Global Assessment Scale (CGAS)

Afterward, volunteers included in the study will complete computer-based Emotion Recognition and Differentiation Tests.

For children exposed to trauma applying to the Istanbul Faculty of Medicine Child and Adolescent Mental Health and Disorders Clinic, psychiatric diagnoses will be shared with their physician upon patient approval. These children will be followed and treated in the clinic according to current guideline-recommended treatment methods.

The planned start date for the study is January 30, 2025, and data analysis will commence afterward. Data will be analyzed using the Statistical Program for Social Sciences (SPSS for Windows, version 21.0). The study is expected to be completed by June 2025.

The coordinating center responsible for the research is the Department of Child and Adolescent Mental Health and Disorders at Istanbul Faculty of Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Having been exposed to at least one traumatic event,
* Being between the ages of 7 and 18,
* The child and/or their parents (or caregivers) having adequate literacy and Turkish communication skills.

Exclusion Criteria:

* The presence of psychotic/manic symptoms in the child or parent during the interview or any condition that makes the interview and assessment impossible (e.g., mental or developmental condition or a different communication language),
* The child or parent refusing to participate in the study,
* The presence of autism spectrum disorder or intellectual disability at a severity that prevents assessment.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients applying to the Child and Adolescent Mental Health and Disorders Outpatient Clinic of Istanbul Faculty of Medicine
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Complex PTSD in Children and Adolescents Exposed to Trauma | Baseline
  The aim of this study is to conduct a psychiatric evaluation of children and adolescents exposed to trauma in the outpatient clinic and to determine the prevalence of PTSD and Complex PTSD (CPTSD) diagnoses.
Examining the Differences Between Groups Who Do Not Have a PTSD Diagnosis, Those Diagnosed with PTSD, and Those Diagnosed with Complex PTSD (CPTSD) | Baseline
  The study aims to compare the clinical characteristics of children exposed to trauma who do not receive a PTSD diagnosis, those diagnosed with PTSD, and those diagnosed with CPTSD, as well as to examine the trauma history of their parents and the severity of their anxiety and depression. Additionally, it will also be examined whether there is a difference in facial emotion recognition skills among these groups.
Adaptation of the International Trauma Questionnaire - Child and Adolescent Version into Turkish and Evaluation of Its Psychometric Properties | Baseline
  Since there is no existing scale in our country to assess CPTSD in children, the study also aims to translate the International Trauma Questionnaire - Child and Adolescent Version into Turkish and evaluate its psychometric properties.

CONTACTS AND LOCATIONS:
Overall Officials: Abdurrahman Cahid Orengul, Associate Professor, MD, Principal Investigator — Istanbul Faculty of Medicine, Child and Adolescent Psychiatry Department
Locations (1):
- Istanbul Faculty of Medicine, Istanbul, Fatih, Turkey (Türkiye)